CLINICAL TRIAL: NCT05285579
Title: Predictive Role of Circulating Biomarkers Involved in Angiogenesis in Metastatic Kidney Cancer in the Era of New Therapeutic Associations: Immunotherapies, Anti-angiogenic
Brief Title: Biomarkers of Angiogenesis for Response to Therapeutic Combination in Advanced or Metastatic Kidney Cancer
Acronym: ANGIOCOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); FONCER contre le cancer (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP211213; IDRCB2021-A02030-41 (Registry Identifier: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Renal Cell Carcinoma; Renal Cancer; Renal Cancer Metastatic
Keywords: renal cell carcinoma; blood biomarkers; predictive factor; tyrosine kinase inhibitor; immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma + tumour tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TKI+ICI: Therapeutic combination tyrosine kinase inhibitor (TKI) + immune checkpoint inhibitors (ICI)
  Interventions: Biological: Blood collection; Other: Tumour samples
- ICI+ICI: Therapeutic combination with different immune checkpoint inhibitors (ICI)
  Interventions: Biological: Blood collection; Other: Tumour samples

INTERVENTIONS:
Biological: Blood collection — Systematic extra blood sampling at inclusion, 6 weeks after inclusion and in case of progression of the cancer
Other: Tumour samples — reuse of tumour tissue collect in usual patient care

SUMMARY:
This is a multicenter, exploratory, prospective study to identify angiogenesis and immune-related biomarkers predictive of progression free survival in patients with metastatic or advanced renal cell carcinoma treated by a combination of immunotherapy and antiangiogenic.

DETAILED DESCRIPTION:
Recently, the management of renal cell carcinoma has undergone major changes with the emergence of combined therapies associating tyrosine kinase inhibitors (TKI) and immune checkpoint inhibitors (ICI) as first line treatments. However, there are no criteria to guide the choice between the different combinations validated and or between ICI combinations. Angiogenesis and immunity are intimately linked and some markers related have could be interesting to predict the efficacy of these combinations. Angiogenesis and immunity are highly related. This link may lead to new biomarkers to be explored to predict the response to TKI + ICI therapy combinations. On this basis, the investigators propose to conduct an open-label exploratory, multicenter prospective trial to study the association between angiogenesis and immune markers and the effect of combined TKI+ICI treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced or metastatic renal carcinoma
* treated in first line with an ICI-ICI or ITK-ICI combination (following current recommendations at inclusion)

Exclusion Criteria:

* Previous systemic treatment for renal cell carcinoma
* Other cancer developed in the last 5 years except local forms apparently healed as basal cell cancer.
* Contraindication for ICI-ICI or TKI-ICI combinations recommended on 1st line
* Refusal to participate in the study
* No affiliation to a social security regime (beneficiary or entitled)
* Vulnerable patients as defined by french law (Public Heath Code sections L1121 -5 to L1121-8) :
* Major patient subjected to legal protection (guardianship, curatorship, protection of justice)
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a metastatic or advanced renal cell carcinoma who will benefit of an ICI-TKI or ICI-ICI combination as a first-line treatment (according to the current guidelines at the time of inclusion).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 24 months
  Time from inclusion to progression documented by imaging and based on RECIST 1.1 and iRECIST criteria or patient death. The iRECIST criteria use the same methods of monitoring tumor lesions as the RECIST 1.1 criteria but a confirmation 4-6 weeks after suspicion of progression is required to confirm or rule out progression because patients undergoing immunotherapy may present pseudo-progressions.

SECONDARY OUTCOMES:
Objective response rate | 24 months
  Observation of a partial or complete response according to RECIST 1.1 criteria during the follow-up
Response duration | 24 months
  Time between the observation of an objective response (partial or complete according to RECIST 1.1 criteria) and the progression

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia MAUGE, PharmD, PhD, Principal Investigator — Assitance Puplique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital européen Georges-Pompidou AP-HP, Paris
  - Hôpital Cochin - AP-HP, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement. Processing of shared data must comply with European General Data Protection Regulation (GDPR).